CLINICAL TRIAL: NCT00273702
Title: An Open-Label Study of N-Acetyl Cysteine in Pathological Gambling
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0511M77412
Record Dates: First submitted 2006-01-06; First posted 2006-01-09 (Estimated); Last update posted 2007-04-30 (Estimated); Status verified 2007-04

CONDITIONS: Pathological Gambling
Keywords: Gambling; Gambler; Gamble; Pathological
MeSH Terms: conditions — Gambling | interventions — Acetylcysteine

INTERVENTIONS:
Drug: N-Acetyl Cysteine

SUMMARY:
After completing all screening evaluations, subjects will receive unblinded N-Acetyl Cysteine 600 mg/day for 2 weeks. The dose will be raised to 1200 mg/day at visit 4 and to 1800 mg/day at visit 6 unless clinical improvement has been attained at a lower dose (clinical improvement will be assessed by the investigator with respect to gambling thoughts, urges and behavior). If it is clinically necessary to modify this schedule (e.g., because of side effects or an adequate response to a lower dose), the dose will be raised more slowly or the target dose will not be reached.

Subjects will start no other psychotropic medications during the study but may continue on previously prescribed psychotropic medications if on a stable dose for 3 months prior to study entry. Psychotherapy of any form (including cognitive-behavioral therapy) will not be initiated during the study but subjects may continue with current psychotherapy if they have been undergoing therapy for at least three months prior to study entry.

Subjects will be evaluated with the PG-YBOCS, G-SAS, CGI, HAM-D, HAM-A and the Sheehan Disability Inventory at screening and at each visit for the remainder of the study. Medication side effects will be evaluated at each study visit. A tablet count will be kept for each dose of medication taken.

DETAILED DESCRIPTION:
Before beginning N-Acetyl Cysteine, all subjects will receive a psychiatric, medical, and family history evaluation as well as the Structured Clinical Interview for DSM-IV (SCID-P) for Axis I disorders. At the screening visit, patients will also receive standard laboratory tests (including ß-HCG), and a physical examination.

The following instruments will be completed at the screening visit and periodically throughout the study: 1) Yale-Brown Obsessive Compulsive Scale Modified for Pathological Gambling (PG-YBOCS), a reliable and valid semi-structured clinician-administered scale that assesses current severity of PG; 2) Gambling Symptom Assessment Scale (G-SAS), a reliable and valid self-report measure of gambling symptoms; 3) the 17-item Hamilton Rating Scale for Depression (HAM-D); 4) the 17-item Hamilton Rating Scale for Anxiety (HAM-A); 5) Clinical Global Impression scale; 6) the Sheehan Disability Inventory; and 7) the Quality of Life Inventory. Safety evaluations, including pulse and blood pressure, and assessment of side effects will be done at each visit.

After completing all screening evaluations, subjects will receive unblinded N-Acetyl Cysteine 600 mg/day for 2 weeks. The dose will be raised to 1200 mg/day at visit 4 and to 1800 mg/day at visit 6 unless clinical improvement has been attained at a lower dose (clinical improvement will be assessed by the investigator with respect to gambling thoughts, urges and behavior). If it is clinically necessary to modify this schedule (e.g., because of side effects or an adequate response to a lower dose), the dose will be raised more slowly or the target dose will not be reached.

Subjects will start no other psychotropic medications during the study but may continue on previously prescribed psychotropic medications if on a stable dose for 3 months prior to study entry. Psychotherapy of any form (including cognitive-behavioral therapy) will not be initiated during the study but subjects may continue with current psychotherapy if they have been undergoing therapy for at least three months prior to study entry.

Subjects will be evaluated with the PG-YBOCS, G-SAS, CGI, HAM-D, HAM-A and the Sheehan Disability Inventory at screening and at each visit for the remainder of the study. Medication side effects will be evaluated at each study visit. A tablet count will be kept for each dose of medication taken.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18-65
* Current DSM-IV PG

Exclusion Criteria:

* Unstable medical illness on physical examination
* History of seizures
* Myocardial infarction within 6 months
* Current pregnancy or lactation, or inadequate contraception in women of childbearing potential
* Clinically significant suicidality
* Lifetime history of DSM-IV bipolar disorder type I, dementia, or schizophrenia or any other DSM-IV psychotic disorder
* Current or recent (past 3 months) DSM-IV substance abuse or dependence
* Illegal substance within 2 weeks of study initiation
* Initiation of psychotherapy or behavior therapy from a mental health professional within 3 months prior to study baseline
* Previous treatment with N-Acetyl Cysteine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-01; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
PG-YBOCS

SECONDARY OUTCOMES:
G-SAS

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, MD, JD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States